CLINICAL TRIAL: NCT02127060
Title: The Effectiveness of Vitamin C in Postoperative Pain Management of Single-level Posterior Lumbar Interbody Fusion (PLIF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Seoul National University, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITC-001
Record Dates: First submitted 2014-04-27; First posted 2014-04-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Fusion of Spine (Disease)
Keywords: vitamin C; effectiveness; pain management; posterior lumbar interbody fusion
MeSH Terms: conditions — Disease; Agnosia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C (Experimental): in postoperative time, vitamin C administered orally with other pain analgesics.
  Interventions: Drug: Vitamin C
- Placebo drug (Placebo Comparator): in postoperative time, vitamin C do not administered.
  Interventions: Drug: Placebo drug

INTERVENTIONS:
Drug: Vitamin C — for 1 month postoperative period, vitamin C was administered orally to the patients.
  Arms: Vitamin C
Drug: Placebo drug — for 1 month postoperative period, placebo medication administered orally to the patients.
  Arms: Placebo drug

SUMMARY:
Postoperative pain management remains a major challenge for surgeons. Despite huge technological advances in pain management, many researchers have documented that unrelieved pain remains common after surgeries, which is estimated that up to 75% of patients do not achieve adequate pain relief postoperatively. The major goal in the management of postoperative pain is to minimize the dose of medications to lessen the side effects while still providing adequate analgesia, because side effects of commonly used pain medications are known to be the reasons that could lead to inadequate postoperative pain treatment. This goal is best accomplished with multimodal analgesia. One agent that can exert antinociceptive and pain reducing effects is vitamin C.

Vitamin C (ascorbic acid) is water-soluble, found throughout the body and is especially highly concentrated in the brain, which has antioxidant and neuroprotective properties. Moreover, it has been proven that the plasma vitamin C concentration decreases after surgery and the requirement for vitamin C increases in surgical patients, possibly due to greater demand caused by increased oxidative stress. Regarding the effect of vitamin C on acute pain, a result from a recent study with the aim to evaluate the potential role of vitamin C in reducing acute pain after laparoscopic cholecystectomy showed that supplementation with oral vitamin C significantly decreased morphine consumption after surgery.

Although vitamin C has potential for relieving postoperative pain, there has not been studied regarding the effectiveness of vitamin C for spine surgery, to date. This trial aimed to evaluate the effectiveness of vitamin C for surgery of lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* patients with a lumbar herniated intervertebral disc, lumbar spondylotic radiculopathy and/or myelopathy, which were diagnosed using lumbar spine radiographs and magnetic resonance images (MRI) that corresponded to clinical manifestations and physical examinations
* patients who underwent one-level PLIF
* patients who volunteered for this study with written consent
* patient who were followed-up for one year or more

Exclusion Criteria:

* fractures, infection, or tumors in the lumbar spine
* patients with hemorrhagic disorders such as hemophilia and thrombocythemia
* patient with a follow-up period of less than one year
* patients who are not suitable for this study judged by the principal investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pain scores on the VAS | Postoperative 1 month
  The pain intensity on lower back and radiating pain to lower extremities were recorded, separately using visual analogue scale (VAS)

SECONDARY OUTCOMES:
Functional outcomes on the ODI and SF-12 | postoperative 3 and12 months
  Postoperative functional outcomes were assessed with Oswestry disability index (ODI) and SF-12 score at postoperative 3 and 12 months.
Union rate | Postoperative 12 months
  fusion outcome was evaluated at postoperative 12 months using dynamic radiographs and CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Jin S. Yeom, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyounggido, South Korea